CLINICAL TRIAL: NCT04836013
Title: Multicenter Randomized Trial of a Combined Probiotic (Lactobacillus Reuteri LMG P-27481 and Lactobacillus Rhamnosus GG (ATCC 53103) for the Prevention of Antibiotic-Associated Diarrhea and Gastrointestinal Symptoms in Children
Brief Title: Combined Lactobacilli (Reuteri LMG P-27481 and GG ATCC 53103) to Prevent Antibiotic Associated Symptoms in Children
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Università degli Studi dell'Insubria (Other)
Responsible Party: Principal Investigator, Silvia Salvatore, Prof. MD, Università degli Studi dell'Insubria
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 52265
Record Dates: First submitted 2021-03-20; First posted 2021-04-08 (Actual); Last update posted 2021-05-04 (Actual); Status verified 2021-05

CONDITIONS: Diarrhea Caused by Drug; Abdominal Pain
Keywords: antibiotics; diarrhea; probiotics; Lactobacillus; children; abdominal pain
MeSH Terms: conditions — Abdominal Pain; Diarrhea

STUDY DESIGN:
Intervention Model Description: Double blind placebo controlled prospective trial
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Double blind trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Probiotic group (Experimental): Lactobacillus reuteri LMG P-27481 and Lactobacillus rhamnosus GG (ATCC 53103), sucralose and isomalt as an oral stick formulation of 1,6 g with a concentration of probiotic of 2x100bilion colony forming unit (CFU) per stick.
  Interventions: Dietary Supplement: combined Lactobacilli
- Placebo group (Placebo Comparator): The placebo will contain 1.6 g per stick of sucralose and isomalt
  Interventions: Other: Placebo

INTERVENTIONS:
Dietary Supplement: combined Lactobacilli — 1 oral stick per day for 30 days starting the day of antibiotic treatment
  Arms: Probiotic group
Other: Placebo — 1 oral stick per day for 30 days starting the day of antibiotic treatment
  Arms: Placebo group

SUMMARY:
This is a prospective multicenter pediatric double-blind, randomized placebo-controlled, parallel group clinical trial intended to evaluate the efficacy, safety and tolerability of a combined probiotic (LGG and L. reuteri LMG P-27481) in the prevention of antibiotic associated diarrhea and gastrointestinal symptoms in hospitalised children treated with antibiotics for proven or suspected bacterial infection.

DETAILED DESCRIPTION:
Eligible children will be randomly assigned to receive the combined probiotic study product (Noos, Roma, Italia)(BCCMTM Bacterial Collection of Ghent, Belgium, Italian Patent: 102016000011071, International Patent Request : PCT/IB 2017/053856), or placebo as additional treatment to the antibiotic therapy. Kind, dose and duration of antibiotic treatment will be decided by the local clinicians according to good medical practice and current recommendations. The first dose of probiotic will be started the same day of starting the antibiotic treatment, immediately after enrollment. Then, each oral stick will be administered orally once daily, in the morning, before breakfast, during the antibiotic treatment and prolonged for 30 days since starting.

Study product The combined probiotic is made by Lactobacillus reuteri LMG P-27481 and Lactobacillus rhamnosus GG (ATCC 53103), sucralose and isomalt as an oral stick formulation of 1.6 g with a concentration of probiotic of 2x1010 colony forming unit (CFU) per stick, launched in the Italian market with the name of Reuterin®GG (Noos, Roma, Italia).

The probiotic and placebo will be prepared centrally by the probiotic producer as identically appearing oral stick. The placebo will contain only sucralose and isomalt, 1.6 g per stick.

Randomization The allocation sequences and randomization lists has been generated by a online computer system. The probiotic -placebo allocation ratio will be of 1:1. To ensure allocation concealment, an independent subject prepared the randomization schedule and sealed envelopes to be sent to the participant centers. Each investigator will control the packaging and labels of trial treatments sent by the producer with a numerical code with no possible identification of the probiotic product compared to the placebo. The allocation will be consecutively assigned for all enrolled subjects. All investigators, participants, and statisticians will be blinded to the assigned treatment throughout the study and during the data analysis. After completing the analysis of the data or in case of sever adverse event the randomization code will be broken and information about the content of the product (probiotic or placebo) will be revealed by the producer, upon the investigator's request.

Monitoring and collection of data At enrollment a standardized form will record age, gender, anthropometric parameters, vital signs, refilling time, site of infection, laboratory tests, kind, dose and route of administration of antibiotic, diet, previous AAD or other gastrointestinal symptoms, comorbidity and associated treatment. Vesikary scale, anthropometric measures, vital signs, refilling time will be also recorded in each patient at enrollment and in case of occurrence of diarrhea. Bristol stool chart will be used to grade the consistency of stools.

Parents or care givers of each children will be instructed to fill in a diary to record the duration of antibiotic treatment and/or other treatment, the intake of the study product, the frequency of daily bowel movements, the consistency of stools (according to the Bristol stool scale), the frequency and intensity (according to a VAS scale, from 0 to 10) of abdominal pain, the presence and duration of fever, vomiting or any other symptoms they considered important, diet changes and general well being (according to a numerical 1-10 scale). The diary will be completed daily for the duration of the probiotic treatment and then weekly till the end of the study. After discharge from the hospital the absence from day care or school, the need of new antibiotic treatment or re-hospitalization will be also noted. In case of diarrhea, fever or other severe symptoms after hospital discharge parents will be instructed to contact the local pediatrician and investigator for clinical evaluation and stool analysis. A clinical visit will be scheduled in all recruited patients after 1, 3 and 6 months from enrollment.

Re-hospitalization will be required in case of severe infection, severe dehydration or whenever considered necessary by clinicians.

Scheduled investigations In all cases presenting diarrhea at least three stool samples will be collected and stool tests will be performed to detect viral, bacterial or C. difficile pathogens. Blood and urine test or radiologial investigations will be decided by the local clinician based on patient's clinical presentation and according to guidelines and good clinical practice.

One additional sample of stools will be collected, whenever possible, in each patient at enrollment, at 1, 3 and 6 months to evaluate fecal calprotectin to indirectly assess intestinal inflammation. In a subgroup of patients (the first 30 recruited in each arms) two other stool samples and a urine sample will be collected and stocked in freezer (-20° C) at the same study point for possible future additional explorative analysis of fecal inflammatory markers (lactoferrine, IgA, IL10 and TNF-α) and metabolomic profile (urine metabolites).

The probiotic producer (Noos S.r.L, Roma, Italia) will gift the probiotic product and placebo for the duration of the study for all children enrolled but has and will have no role in the design and conduct of the study; collection, management, analysis, or interpretation of the data; preparation, review, or approval of the manuscript; or the decision to submit the manuscript for publication. The data of the enrolled subjects will be managed, stored and property of the clinical investigators of the participant centers and of the coordinator center and will be analysed and published anonymously and as aggregate, in the respect of the current legislation on privacy.

ELIGIBILITY:
Inclusion Criteria (all of the following):

* Children aged 12 months to 12 years
* Proven or suspected bacterial infection
* Inpatient children needed antibiotic treatment
* Oral or intravenous or intramuscular antibiotic administration with at least 2 days of duration
* Parental informed consent to the participation to the study

Exclusion Criteria:

* Age below 12 months or above 12 years
* Infections with no or only one day of antibiotic treatment
* Sepsis or severe generalized infection
* Pancreatitis
* Known immunodeficiency or chronic gastrointestinal diseases or heart disease
* Oncologic patients
* Severe neurological impairment or lack of verbal expression
* Enteral or parenteral nutrition
* Gastrointestinal malformations or abdominal surgical interventions
* Central line catheter
* Acute or chronic diarrhea when starting antibiotics
* Current or recent (in the last four weeks) use of any probiotic product
* Antibiotic treatment started earlier than 24 hours before enrollment
* Absence of parental consent

Ages: 12 Months to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 216 (Estimated)
Dates: Start 2021-05-13 (Estimated); Primary Completion 2021-11-30 (Estimated); Study Completion 2022-04-13 (Estimated)

PRIMARY OUTCOMES:
Incidence of antibiotic-associated diarrhea, defined as episodes of otherwise unexplained diarrhea (≥3 loose or liquid stools per day with negative viral and bacterial stool tests), recorded by instructed parents in a structured daily diary. | From the second day after starting antibiotic treatment to 2 weeks after stopping antibiotics
  Both Intention to treat (ITT) and Multivariate linear regression models analysis taking into account age, sex, mode of antibiotic delivery, and the kind of antibiotics and comparison between the two groups will be performed.The relative risk (RR), 95% confidence interval (CI), and number needed to treat (NNT) will also be calculated. The difference between study groups will be considered significant when P-value <0.05 or when the 95% CI for RR will not exceed 1.0.

SECONDARY OUTCOMES:
Number of children with episodes of infective diarrhea; dehydration (by Vesikary scale), fever, abdominal pain, vomiting and constipation (by Bristol stool chart); general well being (by 1-10 scale) as assessed by patient's record form. | 6 months from enrolling
  Instructed parents will record all the above parameters in a structured diary filled daily for the first month and weekly for 5 months. A follow-up evaluation will be done at one month, at 3 and 6 months from enrollment and in cases of diarrhea. The Student's t-test will be used to compare mean values of continuous variables approximating a normal distribution. For non-normally distributed variables, the Mann-Whitney U-test will be used. The chi-square test or Fisher exact test will be used, as appropriate, to compare percentages between the two groups of intervention.

OTHER OUTCOMES:
Number of participants with treatment-related adverse events as assessed by CTCAE v4.0 | From enrolling to all the period of intervention (1 month)
  Participant investigators will record in specific form any adverse event according to CTCAE v4.0
Number of participants with abnormal fecal inflammatory markers (calprotectin, lactoferrine, IgA, IL10 and TNF-α) and urine metabolomic profile | The additional stool and urine sample will be collected at recruitment, after 1 month and after 6 months from enrollment.
  In the first 30 patients recruited an additional stool and urine sample will be collected and stored in freezer (-20°C). Levels of lactoferrine, IgA, IL10 and TNF-α) and metabolomic profile (urine metabolites) will be measured and compared between the two groups.

CONTACTS AND LOCATIONS:
Locations (1):
- Silvia Salvatore, Varese, Italy

IPD SHARING:
Plan to Share IPD: Yes
After publication of the results, upon motivated request
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: From the publication of the study to 5 years
Access Criteria: Mailing to silvia.salvatore@uninsubria.it